CLINICAL TRIAL: NCT00192959
Title: Xenon Inhalation as Cover Sedation During Orthopaedic Surgery in Elderly Subjects Comparing the Effects of Inhaled Xenon and Intravenous Propofol
Brief Title: Xenon Inhalation During Orthopaedic Surgery in Elderly Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Linde AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KF 02-065/03
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-06

CONDITIONS: Anaesthesia; Postoperative Cognitive Function
Keywords: Anaesthesia; Surgery; Postoperative; Neuropsychological test

INTERVENTIONS:
Drug: Xenon vs propofol

SUMMARY:
The primary objective was to explore the feasibility of inhaled xenon for sedation in terms of its effect on postoperative cognitive function in elderly, in comparison with the postoperative cognitive function found after IV propofol sedation in the same population.The secondary objectives were designed to assess the feasibility of xenon sedation in terms of its effects on different neuropsycho-logical test variables, vital signs, sedation levels and safety in elderly orthopaedic subjects.

DETAILED DESCRIPTION:
Primary endpoint: - The primary efficacy parameter was a combined score based on the seven variables derived from four validated neuropsychological tests of cognitive function; Visual Verbal Learning test, Concept Shifting test, Stroop Color Word Interference test and Letter Digit Coding test. The parameter was used for comparing changes in test results between the screening and first postoperative follow-up testing for the treatment groups.Secondary endpoints:- Cognitive performance changes from baseline to the first post-operative follow-up judged separately for each of the seven variables from the changes in the test results.- Cognitive performance changes from baseline to the second postoperative follow-up judged separately and globally for each of the seven variables from the changes in test results.- Adequacy of ventilation (respiratory rate and pulse oximetry)- Adequacy of xenon sedation by monitoring depth of unconsciousness, signs of airway irritation, need for additional sedatives, time to recovery from anaesthesia. - Technical performance of xenon delivery device

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 60 years of age.
* American Soc. of Anaesthesiologists Physical Status Classification (ASA) I-III status [27]
* Referred for elective orthopaedic knee surgery with an anticipated duration of > 45 min
* Expected to remain in hospital for at least 3 days
* Expected to be able to comply with the study protocol throughout the study period
* Mini Mental State Examination (MMSE) score > 23
* Informed consent given

Exclusion Criteria:

* Disease of the CNS (infectious, metabolic, tumours, dementia, epilepsy, major psychiatric disease, confusion/ delirium according to Diagnostic & Statistical Manual of Mental Disorders (DSM) IV criteria)
* Contradiction for spinal anaesthesia
* Contradiction for laryngeal mask
* Regular use of tranquillisers, or antidepressants, if prescribed by psychiatrist for psychosis or depression
* Undergone neuropsychological testing within the last year
* Unable to follow study procedures, illiteracy, or poor comprehension of the language used in the psychometric tests
* Severe visual or auditory disorder
* Alcoholism or drug abuse

CNS disease BMI > 35 Inab

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2004-03; Study Completion 2004-12

PRIMARY OUTCOMES:
Primary endpoint: -cognitive function; Visual Verbal Learning test, Concept Shifting test, Stroop Color Word Interfer

SECONDARY OUTCOMES:
Secondary endpoints:-
Vital signs
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Lars S Rasmussen, MD PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark